CLINICAL TRIAL: NCT05959200
Title: Clinical Performance Evaluation of Two Frequent Replacement Silicone Hydrogel Toric Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CLN109-C001
Record Dates: First submitted 2023-07-13; First posted 2023-07-25 (Actual); Results first posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-10

CONDITIONS: Ametropia; Myopia; Hyperopia; Astigmatism
MeSH Terms: conditions — Refractive Errors; Myopia; Hyperopia; Astigmatism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LID226397, then AOfAHP (Other): Serafilcon A toric contact lenses worn in Period 1, with senofilcon A toric contact lenses worn in Period 2. Each product will be worn bilaterally (in both eyes) during waking hours for approximately 14 days. CLEAR CARE will be used for nightly contact lens cleaning and disinfection.
  Interventions: Device: Serafilcon A toric contact lenses; Device: Senofilcon A toric contact lenses; Device: CLEAR CARE
- AOfAHP, then LID226397 (Other): Senofilcon A toric contact lenses worn in Period 1, with serafilcon A toric contact lenses worn in Period 2. Each product will be worn bilaterally (in both eyes) during waking hours for approximately 14 days. CLEAR CARE will be used for nightly contact lens cleaning and disinfection.
  Interventions: Device: Serafilcon A toric contact lenses; Device: Senofilcon A toric contact lenses; Device: CLEAR CARE

INTERVENTIONS:
Device: Serafilcon A toric contact lenses — Silicone hydrogel contact lenses for the optical correction of refractive ametropia (myopia or hyperopia with astigmatism)
  Other Names: LID226397
Device: Senofilcon A toric contact lenses — Silicone hydrogel contact lenses for the optical correction of refractive ametropia (myopia or hyperopia with astigmatism)
  Other Names: ACUVUE® OASYS for ASTIGMATISM with HYDRACLEAR® PLUS; AOfAHP
Device: CLEAR CARE — Hydrogen peroxide-based contact lens cleaning and disinfecting solution
  Other Names: CLEAR CARE® Cleaning and Disinfecting Solution

SUMMARY:
The primary objective of this study is to evaluate the axis orientation of LID226397 toric contact lenses.

DETAILED DESCRIPTION:
Subjects will be expected to attend 7 visits including a screening visit. The total duration of a subject's participation in the study will be approximately 40 days.

ELIGIBILITY:
Key Inclusion Criteria:

* Successful wearers of any commercial soft toric contact lenses (except AOfAHP and daily disposable lenses) in both eyes with at least 3 months wearing experience, with a minimum wearing time of 5 days per week and 10 hours per day.
* Able to be fit with and wear contact lenses within the available range of sphere & cylinder power and axes.
* Best corrected distance visual acuity greater than or equal to 20/25 Snellen (0.10 logMAR) in each eye as determined by manifest refraction at screening.
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Wearing habitual contact lenses in an extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment.
* Habitual AOfAHP contact lens wearers and habitual daily disposable lens wearers (worn within last 3 months).
* Other exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, CRD Vision Care, Study Director — Alcon Research, LLC
Locations (7):
- United States (7):
  - Dr. Elsa Pao, OD, Oakland, California
  - Pacific Rims Optometry, San Francisco, California
  - Drs. Giedd, P.A., Maitland, Florida
  - Vision Health Institute, Orlando, Florida
  - Franklin Park Eye Center, PC, Franklin Park, Illinois
  - ProCare Vision Centers, Inc., Granville, Ohio
  - Optometry Group, PLLC, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 7 investigative sites located in 1 country (US).
Pre-assignment Details: This reporting group includes all participants exposed to any study lenses evaluated in this study.
Units Other Than Participants: eyes
Groups:
- LID226397, Then AOfAHP: Serafilcon A toric contact lenses worn in Period 1, with senofilcon A toric contact lenses worn in Period 2. Each product was worn bilaterally (in both eyes) during waking hours for approximately 14 days. CLEAR CARE was used for nightly contact lens cleaning and disinfection.
- AOfAHP, Then LID226397: Senofilcon A toric contact lenses worn in Period 1, with serafilcon A toric contact lenses worn in Period 2. Each product was worn bilaterally (in both eyes) during waking hours for approximately 14 days. CLEAR CARE was used for nightly contact lens cleaning and disinfection.
Period: First Wear Period (Approx. 14 Days)
Arm/Group | LID226397, Then AOfAHP | AOfAHP, Then LID226397
Started | 48; 96 eyes | 44; 88 eyes
Completed | 48; 96 eyes | 44; 88 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes
Period: Second Wear Period (Approx. 14 Days)
Arm/Group | LID226397, Then AOfAHP | AOfAHP, Then LID226397
Started | 48; 96 eyes | 44; 88 eyes
Completed | 48; 96 eyes | 44; 88 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: All randomized subjects/eyes exposed to any study lenses evaluated in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | LID226397, Then AOfAHP | AOfAHP, Then LID226397 | Total
Number analyzed (Participants) | 48 | 44 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (9.7) | 32.0 (9.6) | 32.3 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 33 | 55
  Male | 26 | 11 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 35 | 29 | 64
  Black or African American | 2 | 3 | 5
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 10 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 0 | 1 | 1
  Multi-racial | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 10 | 15
  Not Hispanic or Latino | 43 | 33 | 76
  Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Lenses With Axis Orientation Within Plus or Minus 30 Degrees From the Intended Axis at 10 Minutes After Lens Insertion
Description: The investigator will view the contact lens through a slit lamp (biomicroscope) and record the axis orientation (-179° to +180°) as the number of degrees away from the ideal location (90° axis) either positive or negative depending on the direction (nasal [+] or temporal [-]). No hypothesis testing was prespecified for this endpoint.
Time Frame: Day 1 Dispense, 10 minutes after lens insertion, for each wear period. Each wear period is approximately 14 days according to randomization assignment.
Population: Full Analysis Set: All randomized subjects/eyes exposed to any study lenses evaluated in this study.
Measure: Number; unit: percentage of lenses
Units Other Than Participants: eyes
Groups:
- LID226397: Serafilcon A toric contact lenses worn during Period 1 or Period 2, as pre-determined.
- AOfAHP: Senofilcon A toric contact lenses worn during Period 1 or Period 2, as pre-determined.
Arm/Group | LID226397 | AOfAHP
Number analyzed (Participants) | 92 | 92
Number analyzed (eyes) | 184 | 184
percentage of lenses | 100.0 | 100.0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from time of consent to study exit, up to 40 days.
Description: AEs were obtained through solicited and spontaneous comments from subjects and through observations by the investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of subjects. This analysis population includes all subjects/eyes exposed to any study lenses evaluated in this study.
Groups:
- LID226397 Ocular; LID226397 Nonocular: Events reported in this group occurred while exposed to serafilcon A toric contact lenses.
- AOfAHP Ocular; AOfAHP Nonocular: Events reported in this group occurred while exposed to senofilcon A toric contact lenses.
Arm/Group | LID226397 Ocular | LID226397 Nonocular | AOfAHP Ocular | AOfAHP Nonocular
All-Cause Mortality (participants affected / at risk) | 0/184 | 0/92 | 0/184 | 0/92
Serious Adverse Events (participants affected / at risk) | 0/184 | 0/92 | 0/184 | 0/92
Other Adverse Events (participants affected / at risk) | 0/184 | 0/92 | 0/184 | 0/92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study

DOCUMENTS (2):
  • Study Protocol (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT05959200/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-13): https://cdn.clinicaltrials.gov/large-docs/00/NCT05959200/SAP_001.pdf